CLINICAL TRIAL: NCT04381260
Title: RUral dispaRities in prehospitAL STEMI
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00064512
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: ST Elevation Myocardial Infarction; Cardiovascular Diseases
Keywords: cardiovascular emergency; cardiogenic shock
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Cardiovascular Diseases; Shock, Cardiogenic | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 2016-2019 STEMI Registry: Retrospective data will be collected to develop a well-characterized registry of patients treated from 2016-2019 by any of 14 local rural EMS agencies and transported to a facility capable of performing Percutaneous Coronary Intervention. This registry will be used to determine the time to PCI performance for each of the EMS agencies. Time will be adjusted for patient distance from a PCI center using a linear mixed model with a random effect for center and a fixed effect for distance. This process will allow qualitative methods to identify organizational culture, structure, and clinical processes that impact STEMI care from the two highest and lowest performing rural EMS agencies. (n=750)
  Interventions: Other: No intervention
- Key Informant Interviews: After identifying the two highest and lowest performing rural EMS agencies in the 2016-2019 STEMI Registry, key employees from each of those agencies will be recruited to participate in semi-structured key informant interviews. The interviews will assess current clinical care, organizational culture and opportunities for improvement. (n=32)
  Interventions: Other: Interview
- Stakeholder Surveys: Employees at all local EMS agencies will be invited to participate in stakeholder surveys to quantify each agency's use of the care strategies identified during Key Information Interviews. (n=240)
  Interventions: Other: Survey

INTERVENTIONS:
Other: No intervention — There is no intervention for patients included in this group as this is a retrospective data registry only.
  Groups: 2016-2019 STEMI Registry
Other: Interview — Key Informant Interview
  Groups: Key Informant Interviews
Other: Survey — Stakeholder survey
  Groups: Stakeholder Surveys

SUMMARY:
Rural Americans are more likely to be unhealthy, older, living in poverty, uninsured, and medically underserved. The CDC has made achieving health equity and improving cardiovascular health for rural Americans one of their Healthy People 2020 overarching goals. ST-Elevation Myocardial Infarction (STEMI) is a life-threatening cardiovascular emergency that frequently affects people without warning within the communities the Participants live and work. Patients with STEMI have a linear relationship between first medical contact to Percutaneous Coronary Intervention (PCI) time and mortality. Delays are particularly important in STEMI patients with cardiogenic shock, who experience an excess 3.3 deaths per 100 for every 10 minute delay to PCI (for PCI times between 60-180 minutes). Delayed PCI is also associated with a higher rate of long term morbidity, including congestive heart failure and repeat MI. Unfortunately, many rural EMS agencies fail to consistently achieve the recommended 90 minute PCI time goal. Rural agencies are less likely than urban/suburban agencies to meet time goals and this disparity exposes rural patients to excess morbidity and mortality. The American College of Cardiology/American Heart Association (ACC/AHA) endorse the need for prehospital strategies to reduce total ischemic time, particularly in rural settings.

DETAILED DESCRIPTION:
Achieving PCI time goals is influenced by multiple factors, such as patient attributes, agency factors and elements of organizational Emergency Medical Services (EMS) culture. Organizational culture is defined as a set of shared values, beliefs, and assumptions within an organization that influences how people within that organization behave. Differences in organizational culture between hospitals have been associated with both cardiovascular mortality and disease-specific outcomes. Although not yet rigorously studied in the prehospital environment, it is likely that organizational culture contributes to differences in tempo and manner of completing interventions. Prehospital performance accountability and culture have been discussed by experts in EMS magazines but have never been formally studied.

EMS STEMI protocols that include direct transportation to a PCI-capable hospital and pre-hospital PCI center activation improve patient outcomes. Unsuccessful EKG transmission, delayed PCI center activation, and cardiogenic shock have been shown to negatively affect PCI time metrics and patient outcomes. The impact of PCI delays in the rural setting has not been specifically studied. In addition, there are agency-level factors, such as ambulances per capita, number of satellite stations, miles of interstate that likely affect the EMS agency's ability to achieve shorter PCI times for the STEMI patients they care for. This proposal will use mixed methods to identify previously unmeasured components of rural EMS agency organizational culture, structure, care processes, and patient environment that likely influence PCI time and patient outcomes. In addition, this project will identify best practices that can be tested as novel interventions and implemented in rural EMS agencies to improve STEMI time metrics and therefore reduce patient morbidity and mortality.

ELIGIBILITY:
STEMI Registry:

Inclusion:

* Age ≥ 18 years
* Transported to one of four primary PCI centers (Wake Forest Baptist Medical Center (WFBMC), High Point Regional Medical Center (HPRMC), Novant Forsyth Medical Center (FMC), and Moses Cone) by rural agency (county identified rural by 2014 Census) ambulance from 2016-2019
* STEMI identified prior to or upon arrival at hospital

Exclusion:

* None

Key Informant Interviews:

Inclusion:

* Rural agency (county identified rural by 2014 Census)
* Identified as the top or bottom two performing services ranked by overall PCI time by regional STEMI registry patients transported to primary PCI center from 2016-2019
* Hold the position of EMS Director, EMS Medical Director, EMS Training Officer, Paramedic (2), EMT Crew Partner (2) or hold a similar key informant position at a local urban EMS agency (Forsyth county EMS) to allow the interview guide to be field-tested

Exclusion:

* None

Stakeholder Survey:

Inclusion:

* Rural agency (county identified rural by 2014 Census) transported to primary PCI center from 2016-2019
* Hold the position of EMS Director, EMS Medical Director, or EMS Training Officer or be a field provider with a Paramedic or EMT certification

Exclusion:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Registry: Patients included in the registry data will be an all-comers population of patients suffering from STEMI and transported to a primary PCI by one of 14 identified rural EMS agencies between 2016-2019.
  Key Informant Interviews: Participants will be EMS Directors, EMS Medical Directors, EMS Training Officers, Paramedics or EMT Crew Partners at the highest and lowest performing rural EMS agencies as determined by the STEMI registry data.
  Stakeholder Surveys: Survey respondents will be EMS Directors, EMS Medical Directors, EMS Training Officers, Paramedics or EMT Crew Partners at any of the 14 local EMS agencies identified as rural.
Sampling Method: Non-Probability Sample
Enrollment: 473 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Compare the organizational culture, structure, and clinical processes of high and low performing local rural EMS agencies using qualitative methods | 1 day
  Aim 1 will be accomplished by developing a 2016-2019 STEMI data registry, which will be utilized to identify high- and low-performing rural EMS agencies. After identifying these agencies, Key Informants will participate in interviews designed to assess facilitators and barriers to achieving STEMI time metrics.

SECONDARY OUTCOMES:
Quantify the association between factors identified in Aim 1 and PCI time among rural EMS STEMI patient encounters. | 1 day
  Stakeholder surveys will be utilized to quantify each agency's use of factors identified in Aim 1

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Stopyra, MD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.

REFERENCES:
- [Background] Stopyra JP, Miller CD, Hiestand BC, Lefebvre CW, Nicks BA, Cline DM, Askew KL, Riley RF, Russell GB, Burke GL, Herrington D, Hoekstra JW, Mahler SA. Chest Pain Risk Stratification: A Comparison of the 2-Hour Accelerated Diagnostic Protocol (ADAPT) and the HEART Pathway. Crit Pathw Cardiol. 2016 Jun;15(2):46-9. doi: 10.1097/HPC.0000000000000072. PMID 27183253
- [Background] Stopyra JP, Miller CD, Hiestand BC, Lefebvre CW, Nicks BA, Cline DM, Askew KL, Riley RF, Russell GB, Hoekstra JW, Mahler SA. Performance of the EDACS-accelerated Diagnostic Pathway in a Cohort of US Patients with Acute Chest Pain. Crit Pathw Cardiol. 2015 Dec;14(4):134-8. doi: 10.1097/HPC.0000000000000059. PMID 26569652
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX, Anderson JL, Jacobs AK, Halperin JL, Albert NM, Brindis RG, Creager MA, DeMets D, Guyton RA, Hochman JS, Kovacs RJ, Kushner FG, Ohman EM, Stevenson WG, Yancy CW; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2013 Jan 29;127(4):e362-425. doi: 10.1161/CIR.0b013e3182742cf6. Epub 2012 Dec 17. No abstract available. PMID 23247304
- [Background] Armstrong PW, Boden WE. Reperfusion paradox in ST-segment elevation myocardial infarction. Ann Intern Med. 2011 Sep 20;155(6):389-91. doi: 10.7326/0003-4819-155-6-201109200-00008. PMID 21930857
- [Background] Bates ER, Nallamothu BK. Commentary: the role of percutaneous coronary intervention in ST-segment-elevation myocardial infarction. Circulation. 2008 Jul 29;118(5):567-73. doi: 10.1161/CIRCULATIONAHA.108.788620. No abstract available. PMID 18663104
- [Background] Studnek JR, Infinger A, Wilson H, Niess G, Jackson P, Swanson D. Decreased Time from 9-1-1 Call to PCI among Patients Experiencing STEMI Results in a Decreased One Year Mortality. Prehosp Emerg Care. 2018 Nov-Dec;22(6):669-675. doi: 10.1080/10903127.2018.1447621. Epub 2018 Mar 29. PMID 29596009
- [Background] Hsia RY, Shen YC. Percutaneous Coronary Intervention in the United States: Risk Factors for Untimely Access. Health Serv Res. 2016 Apr;51(2):592-609. doi: 10.1111/1475-6773.12335. Epub 2015 Jul 14. PMID 26174998
- [Background] Jollis JG, Al-Khalidi HR, Roettig ML, Berger PB, Corbett CC, Doerfler SM, Fordyce CB, Henry TD, Hollowell L, Magdon-Ismail Z, Kochar A, McCarthy JJ, Monk L, O'Brien P, Rea TD, Shavadia J, Tamis-Holland J, Wilson BH, Ziada KM, Granger CB. Impact of Regionalization of ST-Segment-Elevation Myocardial Infarction Care on Treatment Times and Outcomes for Emergency Medical Services-Transported Patients Presenting to Hospitals With Percutaneous Coronary Intervention: Mission: Lifeline Accelerator-2. Circulation. 2018 Jan 23;137(4):376-387. doi: 10.1161/CIRCULATIONAHA.117.032446. Epub 2017 Nov 14. PMID 29138292
- [Background] Jollis JG, Mehta RH, Roettig ML, Berger PB, Babb JD, Granger CB. Reperfusion of acute myocardial infarction in North Carolina emergency departments (RACE): study design. Am Heart J. 2006 Nov;152(5):851.e1-11. doi: 10.1016/j.ahj.2006.06.036. PMID 17070144
- [Background] Jollis JG, Roettig ML, Aluko AO, Anstrom KJ, Applegate RJ, Babb JD, Berger PB, Bohle DJ, Fletcher SM, Garvey JL, Hathaway WR, Hoekstra JW, Kelly RV, Maddox WT Jr, Shiber JR, Valeri FS, Watling BA, Wilson BH, Granger CB; Reperfusion of Acute Myocardial Infarction in North Carolina Emergency Departments (RACE) Investigators. Implementation of a statewide system for coronary reperfusion for ST-segment elevation myocardial infarction. JAMA. 2007 Nov 28;298(20):2371-80. doi: 10.1001/jama.298.20.joc70124. Epub 2007 Nov 4. PMID 17982184
- [Background] Kragholm K, Lu D, Chiswell K, Al-Khalidi HR, Roettig ML, Roe M, Jollis J, Granger CB. Improvement in Care and Outcomes for Emergency Medical Service-Transported Patients With ST-Elevation Myocardial Infarction (STEMI) With and Without Prehospital Cardiac Arrest: A Mission: Lifeline STEMI Accelerator Study. J Am Heart Assoc. 2017 Oct 11;6(10):e005717. doi: 10.1161/JAHA.117.005717. PMID 29021273
- [Background] Jollis JG, Al-Khalidi HR, Roettig ML, Berger PB, Corbett CC, Dauerman HL, Fordyce CB, Fox K, Garvey JL, Gregory T, Henry TD, Rokos IC, Sherwood MW, Suter RE, Wilson BH, Granger CB; Mission: Lifeline STEMI Systems Accelerator Project. Regional Systems of Care Demonstration Project: American Heart Association Mission: Lifeline STEMI Systems Accelerator. Circulation. 2016 Aug 2;134(5):365-74. doi: 10.1161/CIRCULATIONAHA.115.019474. PMID 27482000
- [Background] Bagai A, Al-Khalidi HR, Sherwood MW, Munoz D, Roettig ML, Jollis JG, Granger CB. Regional systems of care demonstration project: Mission: Lifeline STEMI Systems Accelerator: design and methodology. Am Heart J. 2014 Jan;167(1):15-21.e3. doi: 10.1016/j.ahj.2013.10.005. Epub 2013 Oct 23. PMID 24332137
- [Background] Steinberg BA, Jollis JG, Winkler A, Granger C, Newby LK. Treatment pathways and quality improvement for patients with acute myocardial infarction at a tertiary care center. Crit Pathw Cardiol. 2012 Jun;11(2):77-80. doi: 10.1097/HPC.0b013e318252990c. PMID 22595818
- [Background] Fordyce CB, Al-Khalidi HR, Jollis JG, Roettig ML, Gu J, Bagai A, Berger PB, Corbett CC, Dauerman HL, Fox K, Garvey JL, Henry TD, Rokos IC, Sherwood MW, Wilson BH, Granger CB; STEMI Systems Accelerator Project. Association of Rapid Care Process Implementation on Reperfusion Times Across Multiple ST-Segment-Elevation Myocardial Infarction Networks. Circ Cardiovasc Interv. 2017 Jan;10(1):e004061. doi: 10.1161/CIRCINTERVENTIONS.116.004061. PMID 28082714
- [Background] Jollis JG, Al-Khalidi HR, Monk L, Roettig ML, Garvey JL, Aluko AO, Wilson BH, Applegate RJ, Mears G, Corbett CC, Granger CB; Regional Approach to Cardiovascular Emergencies (RACE) Investigators. Expansion of a regional ST-segment-elevation myocardial infarction system to an entire state. Circulation. 2012 Jul 10;126(2):189-95. doi: 10.1161/CIRCULATIONAHA.111.068049. Epub 2012 Jun 4. PMID 22665718
- [Background] Bagai A, Al-Khalidi HR, Munoz D, Monk L, Roettig ML, Corbett CC, Garvey JL, Wilson BH, Granger CB, Jollis JG. Bypassing the emergency department and time to reperfusion in patients with prehospital ST-segment-elevation: findings from the reperfusion in acute myocardial infarction in Carolina Emergency Departments project. Circ Cardiovasc Interv. 2013 Aug;6(4):399-406. doi: 10.1161/CIRCINTERVENTIONS.112.000136. Epub 2013 Jul 16. PMID 23861465
- [Background] Rasmussen DK, Washington A, Dougherty J, Fetcko L. Door-to-balloon time for primary percutaneous coronary intervention: how does Northern West Virginia compare? J Emerg Med. 2012 Sep;43(3):413-6. doi: 10.1016/j.jemermed.2011.06.050. Epub 2011 Oct 26. PMID 22032813
- [Background] Blankenship JC, Scott TD, Skelding KA, Haldis TA, Tompkins-Weber K, Sledgen MY, Donegan MA, Buckley JW, Sartorius JA, Hodgson JM, Berger PB. Door-to-balloon times under 90 min can be routinely achieved for patients transferred for ST-segment elevation myocardial infarction percutaneous coronary intervention in a rural setting. J Am Coll Cardiol. 2011 Jan 18;57(3):272-9. doi: 10.1016/j.jacc.2010.06.056. PMID 21232663
- [Background] Abrams TE, Vaughan-Sarrazin M, Kaboli PJ. Mortality and revascularization following admission for acute myocardial infarction: implication for rural veterans. J Rural Health. 2010 Fall;26(4):310-7. doi: 10.1111/j.1748-0361.2010.00318.x. Epub 2010 Aug 17. PMID 21029165
- [Background] James CV, Moonesinghe R, Wilson-Frederick SM, Hall JE, Penman-Aguilar A, Bouye K. Racial/Ethnic Health Disparities Among Rural Adults-United States, 2012-2015: MMWR Surveillance Summaries / November 17, 2017 / 66(23);1-9. J Health Care Poor Underserved. 2018;29(1):19-34. doi: 10.1353/hpu.2018.0003. PMID 29503284
- [Background] Nam J, Caners K, Bowen JM, Welsford M, O'Reilly D. Systematic review and meta-analysis of the benefits of out-of-hospital 12-lead ECG and advance notification in ST-segment elevation myocardial infarction patients. Ann Emerg Med. 2014 Aug;64(2):176-86, 186.e1-9. doi: 10.1016/j.annemergmed.2013.11.016. Epub 2013 Dec 22. PMID 24368054
- [Background] Savage ML, Poon KK, Johnston EM, Raffel OC, Incani A, Bryant J, Rashford S, Pincus M, Walters DL. Pre-hospital ambulance notification and initiation of treatment of ST elevation myocardial infarction is associated with significant reduction in door-to-balloon time for primary PCI. Heart Lung Circ. 2014 May;23(5):435-43. doi: 10.1016/j.hlc.2013.11.015. Epub 2013 Dec 11. PMID 24388497
- [Background] Quinn T, Johnsen S, Gale CP, Snooks H, McLean S, Woollard M, Weston C; Myocardial Ischaemia National Audit Project (MINAP) Steering Group. Effects of prehospital 12-lead ECG on processes of care and mortality in acute coronary syndrome: a linked cohort study from the Myocardial Ischaemia National Audit Project. Heart. 2014 Jun;100(12):944-50. doi: 10.1136/heartjnl-2013-304599. Epub 2014 Apr 14. PMID 24732676
- [Background] Foo CY, Bonsu KO, Nallamothu BK, Reid CM, Dhippayom T, Reidpath DD, Chaiyakunapruk N. Coronary intervention door-to-balloon time and outcomes in ST-elevation myocardial infarction: a meta-analysis. Heart. 2018 Aug;104(16):1362-1369. doi: 10.1136/heartjnl-2017-312517. Epub 2018 Feb 5. PMID 29437704
- [Background] Stopyra JP, Courage C, Davis CA, Hiestand BC, Nelson RD, Winslow JE. Impact of a "Team-focused CPR" Protocol on Out-of-hospital Cardiac Arrest Survival in a Rural EMS System. Crit Pathw Cardiol. 2016 Sep;15(3):98-102. doi: 10.1097/HPC.0000000000000080. PMID 27465004
- [Background] Stopyra JP, Harper WS, Higgins TJ, Prokesova JV, Winslow JE, Nelson RD, Alson RL, Davis CA, Russell GB, Miller CD, Mahler SA. Prehospital Modified HEART Score Predictive of 30-Day Adverse Cardiac Events. Prehosp Disaster Med. 2018 Feb;33(1):58-62. doi: 10.1017/S1049023X17007154. Epub 2018 Jan 10. PMID 29316995
- [Background] Mell HK, Mumma SN, Hiestand B, Carr BG, Holland T, Stopyra J. Emergency Medical Services Response Times in Rural, Suburban, and Urban Areas. JAMA Surg. 2017 Oct 1;152(10):983-984. doi: 10.1001/jamasurg.2017.2230. PMID 28724118
- [Background] Scholz KH, Maier SKG, Maier LS, Lengenfelder B, Jacobshagen C, Jung J, Fleischmann C, Werner GS, Olbrich HG, Ott R, Mudra H, Seidl K, Schulze PC, Weiss C, Haimerl J, Friede T, Meyer T. Impact of treatment delay on mortality in ST-segment elevation myocardial infarction (STEMI) patients presenting with and without haemodynamic instability: results from the German prospective, multicentre FITT-STEMI trial. Eur Heart J. 2018 Apr 1;39(13):1065-1074. doi: 10.1093/eurheartj/ehy004. PMID 29452351
- [Background] Terkelsen CJ, Sorensen JT, Maeng M, Jensen LO, Tilsted HH, Trautner S, Vach W, Johnsen SP, Thuesen L, Lassen JF. System delay and mortality among patients with STEMI treated with primary percutaneous coronary intervention. JAMA. 2010 Aug 18;304(7):763-71. doi: 10.1001/jama.2010.1139. PMID 20716739
- [Background] Terkelsen CJ, Jensen LO, Tilsted HH, Trautner S, Johnsen SP, Vach W, Botker HE, Thuesen L, Lassen JF. Health care system delay and heart failure in patients with ST-segment elevation myocardial infarction treated with primary percutaneous coronary intervention: follow-up of population-based medical registry data. Ann Intern Med. 2011 Sep 20;155(6):361-7. doi: 10.7326/0003-4819-155-6-201109200-00004. PMID 21930853
- [Background] Lambert L, Brown K, Segal E, Brophy J, Rodes-Cabau J, Bogaty P. Association between timeliness of reperfusion therapy and clinical outcomes in ST-elevation myocardial infarction. JAMA. 2010 Jun 2;303(21):2148-55. doi: 10.1001/jama.2010.712. PMID 20516415
- [Background] Bennin CK, Ibrahim S, Al-Saffar F, Box LC, Strom JA. Achieving timely percutaneous reperfusion for rural ST-elevation myocardial infarction patients by direct transport to an urban PCI-hospital. J Geriatr Cardiol. 2016 Oct;13(10):840-845. doi: 10.11909/j.issn.1671-5411.2016.10.012. PMID 27928226
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; American College of Emergency Physicians; Society for Cardiovascular Angiography and Interventions. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines: developed in collaboration with the American College of Emergency Physicians and Society for Cardiovascular Angiography and Interventions. Catheter Cardiovasc Interv. 2013 Jul 1;82(1):E1-27. doi: 10.1002/ccd.24776. Epub 2013 Jan 8. No abstract available. PMID 23299937
- [Background] Dauerman HL, Bates ER, Kontos MC, Li S, Garvey JL, Henry TD, Manoukian SV, Roe MT. Nationwide Analysis of Patients With ST-Segment-Elevation Myocardial Infarction Transferred for Primary Percutaneous Intervention: Findings From the American Heart Association Mission: Lifeline Program. Circ Cardiovasc Interv. 2015 May;8(5):e002450. doi: 10.1161/CIRCINTERVENTIONS.114.002450. PMID 25901044
- [Background] Langabeer JR 2nd, Prasad S, Seo M, Smith DT, Segrest W, Owan T, Gerard D, Eisenhauer MD. The effect of interhospital transfers, emergency medical services, and distance on ischemic time in a rural ST-elevation myocardial infarction system of care. Am J Emerg Med. 2015 Jul;33(7):913-6. doi: 10.1016/j.ajem.2015.04.009. Epub 2015 Apr 10. PMID 25910668
- [Background] Rhudy JP Jr, Alexandrov AW, Hyrkas KE, Jablonski-Jaudon RA, Pryor ER, Wang HE, Bakitas MA. Geographic access to interventional cardiology services in one rural state. Heart Lung. 2016 Sep-Oct;45(5):434-40. doi: 10.1016/j.hrtlng.2016.07.002. Epub 2016 Aug 1. PMID 27493022
- [Background] Tanguay A, Dallaire R, Hebert D, Begin F, Fleet R. Rural Patient Access to Primary Percutaneous Coronary Intervention Centers is Improved by a Novel Integrated Telemedicine Prehospital System. J Emerg Med. 2015 Nov;49(5):657-64. doi: 10.1016/j.jemermed.2015.05.009. Epub 2015 Jul 26. PMID 26215451
- [Background] Ravasi D SM. Responding to Organizatinal Identity Threats: Exploring the Role of Organizational Culture. The Academy of Management Journal 2006;49:433-58.
- [Background] Webster TR, Curry L, Berg D, Radford M, Krumholz HM, Bradley EH. Organizational resiliency: how top-performing hospitals respond to setbacks in improving quality of cardiac care. J Healthc Manag. 2008 May-Jun;53(3):169-81; discussion 181-2. PMID 18546919
- [Background] Bradley EH, Curry LA, Spatz ES, Herrin J, Cherlin EJ, Curtis JP, Thompson JW, Ting HH, Wang Y, Krumholz HM. Hospital strategies for reducing risk-standardized mortality rates in acute myocardial infarction. Ann Intern Med. 2012 May 1;156(9):618-26. doi: 10.7326/0003-4819-156-9-201205010-00003. PMID 22547471
- [Background] Bradley EH, Curry LA, Webster TR, Mattera JA, Roumanis SA, Radford MJ, McNamara RL, Barton BA, Berg DN, Krumholz HM. Achieving rapid door-to-balloon times: how top hospitals improve complex clinical systems. Circulation. 2006 Feb 28;113(8):1079-85. doi: 10.1161/CIRCULATIONAHA.105.590133. Epub 2006 Feb 20. PMID 16490818
- [Background] Bradley EH, Roumanis SA, Radford MJ, Webster TR, McNamara RL, Mattera JA, Barton BA, Berg DN, Portnay EL, Moscovitz H, Parkosewich J, Holmboe ES, Blaney M, Krumholz HM. Achieving door-to-balloon times that meet quality guidelines: how do successful hospitals do it? J Am Coll Cardiol. 2005 Oct 4;46(7):1236-41. doi: 10.1016/j.jacc.2005.07.009. PMID 16198837
- [Background] Curry LA, Spatz E, Cherlin E, Thompson JW, Berg D, Ting HH, Decker C, Krumholz HM, Bradley EH. What distinguishes top-performing hospitals in acute myocardial infarction mortality rates? A qualitative study. Ann Intern Med. 2011 Mar 15;154(6):384-90. doi: 10.7326/0003-4819-154-6-201103150-00003. PMID 21403074
- [Background] Brunetti ND, Dellegrottaglie G, Lopriore C, Di Giuseppe G, De Gennaro L, Lanzone S, Di Biase M. Prehospital telemedicine electrocardiogram triage for a regional public emergency medical service: is it worth it? A preliminary cost analysis. Clin Cardiol. 2014 Mar;37(3):140-5. doi: 10.1002/clc.22234. Epub 2014 Jan 22. PMID 24452666
- [Background] Rasmussen MB, Frost L, Stengaard C, Brorholt-Petersen JU, Dodt KK, Sondergaard HM, Terkelsen CJ. Diagnostic performance and system delay using telemedicine for prehospital diagnosis in triaging and treatment of STEMI. Heart. 2014 May;100(9):711-5. doi: 10.1136/heartjnl-2013-304576. Epub 2014 Mar 17. PMID 24637516
- [Background] Sorensen JT, Terkelsen CJ, Norgaard BL, Trautner S, Hansen TM, Botker HE, Lassen JF, Andersen HR. Urban and rural implementation of pre-hospital diagnosis and direct referral for primary percutaneous coronary intervention in patients with acute ST-elevation myocardial infarction. Eur Heart J. 2011 Feb;32(4):430-6. doi: 10.1093/eurheartj/ehq437. Epub 2010 Dec 7. PMID 21138933
- [Background] D'Arcy NT, Bosson N, Kaji AH, Bui QT, French WJ, Thomas JL, Elizarraraz Y, Gonzalez N, Garcia J, Niemann JT. Weekly Checks Improve Real-Time Prehospital ECG Transmission in Suspected STEMI. Prehosp Disaster Med. 2018 Jun;33(3):245-249. doi: 10.1017/S1049023X18000341. Epub 2018 Apr 30. PMID 29708085
- [Background] Roswell RO, Greet B, Parikh P, Mignatti A, Freese J, Lobach I, Guo Y, Keller N, Radford M, Bangalore S. From door-to-balloon time to contact-to-device time: predictors of achieving target times in patients with ST-elevation myocardial infarction. Clin Cardiol. 2014 Jul;37(7):389-94. doi: 10.1002/clc.22278. Epub 2014 Apr 3. PMID 24700343
- [Background] Bradley EH, Curry LA, Ramanadhan S, Rowe L, Nembhard IM, Krumholz HM. Research in action: using positive deviance to improve quality of health care. Implement Sci. 2009 May 8;4:25. doi: 10.1186/1748-5908-4-25. PMID 19426507
- [Background] Bandura A. Social Foundations of Thought and Action: A Social Cognitive Theory. 1986.
- [Background] Colorafi KJ, Evans B. Qualitative Descriptive Methods in Health Science Research. HERD. 2016 Jul;9(4):16-25. doi: 10.1177/1937586715614171. Epub 2016 Jan 19. PMID 26791375
- [Background] Grossoehme DH. Overview of qualitative research. J Health Care Chaplain. 2014;20(3):109-22. doi: 10.1080/08854726.2014.925660. PMID 24926897
- [Background] Luft HS. Data and methods to facilitate delivery system reform: harnessing collective intelligence to learn from positive deviance. Health Serv Res. 2010 Oct;45(5 Pt 2):1570-80. doi: 10.1111/j.1475-6773.2010.01148.x. Epub 2010 Aug 2. PMID 21054373
- [Background] Boulkedid R, Abdoul H, Loustau M, Sibony O, Alberti C. Using and reporting the Delphi method for selecting healthcare quality indicators: a systematic review. PLoS One. 2011;6(6):e20476. doi: 10.1371/journal.pone.0020476. Epub 2011 Jun 9. PMID 21694759
- [Background] Hsu C-CS, Brian A. The Delphi Technique: Making Sense of Consensus. Practical Assessment Research & Evaluation 2007;12:1-7.
- [Background] Lynn MR. Determination and quantification of content validity. Nurs Res. 1986 Nov-Dec;35(6):382-5. No abstract available. PMID 3640358